CLINICAL TRIAL: NCT01404806
Title: A Phase 1, Open Label, Study in Healthy Female Subjects to Describe GSK1349572 Exposure in Blood, Cervicovaginal Fluid, and Cervical and Vaginal Tissue Following Single and Multiple Dosing of GSK1349572
Brief Title: GSK1349572 Exposure in Blood, Cervicovaginal Fluid, and Cervical and Vaginal Tissue in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Kristine Patterson, MD, Physician, Division of Infectious Disease, University of North Carolina, Chapel Hill
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 11-1011
Record Dates: First submitted 2011-07-25; First posted 2011-07-28 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Adult Females
MeSH Terms: interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK1349572 (Experimental)
  Interventions: Drug: GSK1349572 (dolutegravir)

INTERVENTIONS:
Drug: GSK1349572 (dolutegravir) — Subjects will take an oral daily 50mg dose of GSK1349572 for 5-7 days. GSK1349572 in the CVF and BP will be measured over 24 hours after both the initial dose, and once steady state is reached 5-7 days later at the following time points: 0 (pre-dose) 1, 2, 3, 4, 5, 6, 8, 12, 18, and 24h. Cervical and vaginal biopsies will be collected once at initial dose at either 3, 6, 12 or 24 hours post dose, and again at steady state at the same single time point. Samples will be collected from 2 subjects per time point. BP and CVF samples will be obtained at 48 and 72 hours following the final GSK1349572 dose.

SUMMARY:
The purpose of this study is to describe drug concentrations of an investigational HIV medication, GSK1349572, in blood plasma, cervicovaginal fluid, vaginal and cervical tissue in HIV negative women.

DETAILED DESCRIPTION:
Purpose: The purpose of this study is to describe first dose and steady state pharmacokinetics of GSK1349572 in cervicovaginal fluid (CVF) and vaginal (VT) and cervical (CT) tissue compared to blood plasma (BP) in HIV-1 negative women. Based on current literature, GSK1349572 has demonstrated a desirable pharmacokinetic profile in BP, including low to moderate pharmacokinetic variability (CV% 9-41), extended t1/2 (13-15h) and trough concentrations which remain 25-fold higher than the protein-adjusted IC90 ~0.064µg/mL for wild type virus. Understanding pharmacokinetic behavior of GSK1349572 in multiple female biological compartments will inform its role in sterilizing the genital tract in HIV-infected women, as well as protect mucosal tissue against HIV infection (pre/post-exposure prophylaxis).

ELIGIBILITY:
Inclusion Criteria:

* Healthy pre-menopausal female subjects between the ages of 18 and 35 years, inclusive, with an intact uterus and cervix.
* Body Mass Index (BMI) of approximately 18-30 kg/m2 and a total body weight of >50kg (110 lbs)
* Negative serum pregnancy test at screening and should be using at least one of the following methods of contraception:

  1. Abstinence
  2. Bilateral tubal ligation
  3. Condom with spermicidal gel or foam
  4. Stable male partner who has had a vasectomy, or stable female only partners
  5. Hormonal contraceptives (oral) provided the subject remains on the treatment until the follow-up visit and has been using oral contraceptives for at least 3 months prior to the first dose of trial medication
* Must agree to abstain from use of intravaginal products for 72 hours prior to the screening visit
* Must agree to abstain from any sexual activity for 72 hours prior to the Day 1 study visit and through study completion
* Previous gynecological examination with documentation of a normal Pap smear within the last year as part of clinical care
* Regular menstrual cycles with at least 21 days between menses (unless on contraception that causes amenorrhea or irregular menses)

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
* History of hysterectomy, loop electrosurgical excision procedure (LEEP), conization or cryosurgery
* Pregnant or lactating
* Unwilling to refrain from sexual intercourse or from using intra-vaginal medications/products from 72 hours prior to Day 1 until discharge from the study
* Any condition possibly affecting drug absorption (eg, gastrectomy)
* Positive urine drug screen
* Active hepatitis B infection
* Active hepatitis C infection
* A positive test for bacterial vaginosis, syphilis, gonorrhea, chlamydia, HIV, HSV-2 (active lesions) or trichomonas at screening
* History of regular use of tobacco- or nicotine-containing products exceeding 5 cigarettes per day within 3 months prior to screening
* History of regular alcohol consumption exceeding 14 drinks [1 drink = 5 ounces (150mL)] of wine or 12 ounces (360mL) of beer or 1.5 ounces (45mL) of spirits per week
* History of bleeding or clotting disorders
* Documented allergic reaction to lidocaine, silver nitrate, ferric subsulfate solution (Monsel's solution) or any iron containing products.
* Treatment with an investigational drug within 4 months preceding the first dose of trial medication.
* Use of clinically significant prescription or non-prescription drugs within 7 days prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Blood donation of approximately 1 pint (500mL) within 56 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Unwilling to abstain from alcohol use from 48 hours prior to the first dose of study medication until after the follow-up visit.
* Using an intrauterine device for contraception.
* Using depo-medroxyprogesterone (DepoProvera®) for contraception.
* Systolic blood pressure is outside the range of 90-140mmHg, diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100 bpm for female subjects even after a single repeat reading.
* Any clinically significant abnormalities to pulse or conduction observed on screening ECG

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Area under the concentration time curve in blood plasma after a single dose | 24 hours
  The area under the concentration time curve will be determined from all sample collection time points over a 24 hour period for blood plasma. Sample collection will occur pre-dose, then 1, 2, 3, 4, 5, 6, 8, 12, 18, and 24 hours post-dose. AUCs will be determined for individual subjects and for all subjects combined.
Peak Concentration (Cmax) after a single dose in blood plasma | 24 hours
  Peak drug concentrations in blood plasma will be determine from samples taken pre-dose, then at 1, 2, 3, 4, 5, 6, 8, 12, 18, and 24 hours post-dose after a first dose in each subject and across all subjects
Area under the concentration time curve in cervicovaginal fluid after a single dose | 24 hours
  The area under the concentration time curve will be determined from all sample collection time points over a 24 hour period for cervicovaginal fluid. Sample collection will occur pre-dose, then 1, 2, 3, 4, 5, 6, 8, 12, 18, and 24 hours post-dose. AUCs will be determined for individual subjects and for all subjects combined.
Area under the concentration time curve in cervical and vaginal tissue after a single dose | 24 hours
  The area under the concentration time curve will be determined from all sample collection time points over a 24 hour period for cervical and vaginal tissue samples. Sample collection will occur at one time point per subject, either at 3, 6, 12, or 24 hours post-dose. AUCs will be determined for all subjects combined.
Peak Concentration (Cmax) after a single dose in cervicovaginal fluid | 24 hours
  Peak drug concentrations in cervicovaginal fluid will be determine from samples taken pre-dose, then at 1, 2, 3, 4, 5, 6, 8, 12, 18, and 24 hours post-dose after a first dose in each subject and across all subjects
Peak Concentration (Cmax) after a single dose in cervical and vaginal tissue | 24 hours
  Peak drug concentrations in cervical and vaginal tissue will be determine from samples taken at one time point per subject at either 3, 6, 12, or 24 hours post-dose after a first dose across all subjects
Area under the concentration time curve for cervicovaginal fluid at steady state | 72 hours
  The area under the concentration time curve will be determined from all sample collection time points over a 72 hour period for cervicovaginal fluid after steady state is reached. Sample collection will occur pre-dose, then at 1, 2, 3, 4, 5, 6, 8, 12, 18, 24, 48, and 72 hours post-dose.
Area under the concentration time curve in cervical and vaginal tissue at steady state | 24 hours
  The area under the concentration time curve will be determined from all sample collection time points over a 24 hour period for cervical/vaginal tissue after steady state is reached. Sample collection will occur at one time point per subject, either 3, 6, 12 or 24 hours post dose and the combined data from all subjects will be used to determine the AUC.
Peak concentration (Cmax) in cervicovaginal fluid at steady state | 72 hours
  Peak drug concentrations in cervicovaginal fluid will be determined at steady state in each subject and across all subjects. Samples will be collected pre-dose, then at 1, 2, 3, 4, 5, 6, 8, 12, 18, 24, 48, and 72 hours post-dose.
Peak concentration (Cmax) in blood plasma at steady state | 24 hours
  Peak drug concentrations in cervical/vaginal tissue will be determined at steady state. Each subject will have samples collected at one time point, either 3, 6, 12, or 24 hours post-dose and the peak will be determined by the combined data of all subjects
Area under the concentration time curve in blood plasma at steady state | 72 hours
  The area under the concentration time curve will be determined from all sample collection time points over a 72 hour period for blood plasma. Sample collection will occur pre-dose, then 1, 2, 3, 4, 5, 6, 8, 12, 18, 24, 48, and 72 hours post-dose. AUCs will be determined for individual subjects and for all subjects combined.
Peak concentration (Cmax) in blood plasma at steady state | 72 hours
  Peak drug concentrations in blood plasma will be determined at steady state in each subject and across all subjects. Samples will be collected pre-dose, then at 1, 2, 3, 4, 5, 6, 8, 12, 18, 24, 48, and 72 hours post-dose.
Area under the concentration time curve ratios after a single dose | 24 hours
  AUC ratios will be determined to compare blood plasma concentrations after a single dose with concentrations in cervicovaginal and cervical and vaginal tissues.
Area under the concentration time curve ratios at steady state | 72 hours
  AUC ratios will be determined to compare concentrations in cervicovaginal fluid and tissues to blood plasma concentrations at steady state.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine B. Patterson, M.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Adams JL, Patterson KB, Prince HM, Sykes C, Greener BN, Dumond JB, Kashuba AD. Single and multiple dose pharmacokinetics of dolutegravir in the genital tract of HIV-negative women. Antivir Ther. 2013;18(8):1005-13. doi: 10.3851/IMP2665. Epub 2013 Jul 31. PMID 23899439